CLINICAL TRIAL: NCT04680676
Title: A Phase II, Randomised, Double-blind, Placebo-controlled, Parallel-group, Dose-ranging, Proof-of-concept Trial of BI 730357 Given for 12 Weeks in Patients With Active Psoriatic Arthritis
Brief Title: A Study to Test Different Doses of BI 730357 and Find Out Whether They Reduce Symptoms in People With Active Psoriatic Arthritis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Program discontinued
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1407-0004; 2019-003182-17 (EudraCT Number)
Record Dates: First submitted 2020-11-13; First posted 2020-12-23 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Arthritis, Psoriatic
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BI 730357 - low dose (Experimental)
  Interventions: Drug: BI 730357
- BI 730357 - medium dose (Experimental)
  Interventions: Drug: BI 730357
- BI 730357 - high dose (Experimental)
  Interventions: Drug: BI 730357
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 730357 — BI 730357
  Arms: BI 730357 - high dose; BI 730357 - low dose; BI 730357 - medium dose
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is open to adults with active psoriatic arthritis who have tender and swollen joints. The purpose of this study is to find out whether a medicine called BI 730357 helps to reduce symptoms and to prevent damage to joints.

Three different doses of BI 730357 are tested. Participants are put into 4 groups by chance. Participants in 3 of the 4 groups take BI 730357. Participants in the fourth group take placebo. Participants take BI 730357 or placebo as tablets once a day. Placebo tablets look like BI 730357 tablets but do not contain any medicine.

Participants are in the study for about 4.5 months. During this time, they visit the study site about 8 times. At these visits, doctors check whether the swelling of inflamed joints has changed. The results between the BI 730357 and placebo groups are then compared. Doctors also regularly check the general health of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18* years and ≤ 75 years at screening, males or females

  -- Except in countries where the minimum age of consent is greater than 18, in which case the minimum age is the minimum age of consent.
* Signed and dated written informed consent in accordance with International Conference on Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Have Psoriatic Arthritis (PsA) symptoms for ≥ 6 months prior to screening, as assessed by the investigator
* Have PsA on the basis of the Classification Criteria for Psoriatic Arthritis (CASPAR) with peripheral symptoms at screening visit, as assessed by the investigator
* Have ≥ 3 tender joints and ≥ 3 swollen joints at screening and randomisation visits, as assessed by the investigator
* At least one Psoriasis (PsO) skin or nail lesion or a documented personal history of PsO at screening, as assessed by the investigator
* If patients receive concurrent PsA treatments, these need to be on stable doses as below:

  * For patients receiving Methotrexate (MTX): patient has received treatment for ≥ 3 months, with stable dose and stable route of administration for ≥ 4 weeks prior to randomisation to End Of Observation (EOO); patients on MTX should be taking folic acid supplementation according to local standard of care before randomisation and during the trial to minimize the likelihood of MTX associated toxicity
  * For patients receiving oral corticosteroids: the patient must be on a stable dose for ≥ 2 weeks prior to randomisation to EOO
  * For patients receiving non-steroidal anti-inflammatory drugs (NSAIDs) or paracetamol/acetaminophen Pro re nata (PRN): the patient must be on stable dose for ≥ 2 weeks prior to randomisation to EOO
* Women of child-bearing potential (A woman is considered of childbearing potential, i.e., fertile, following menarche and until becoming postmenopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. Tubal ligation is NOT a method of permanent sterilisation. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.) must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. Such methods should be used throughout the study and the patient must agree to periodic pregnancy testing during participation in the trial. There are no specific contraceptive requirements for male participants.

Patients (males or females) following the national regulatory guidelines regarding contraception if receiving MTX as background therapy.

Exclusion Criteria:

* Major chronic inflammatory or connective tissue disease other than PsA (e.g. rheumatoid arthritis, systemic lupus erythematosus, ankylosing spondylitis, Lyme disease, gout) or fibromyalgia, as assessed by the investigator
* Active uveitis or uveitis within 4 weeks prior to randomisation, assessed by the investigator
* Suspected or diagnosed inflammatory bowel disease, assessed by the investigator
* Previous exposure to BI 730357
* Prior use of any therapeutic agent directly targeted to Interleukin (IL)-12/23, IL-23 or IL-17
* Prior use of more than two different Tumor necrosis factor inhibitor (TNFi) agents
* Use of the following treatments:

  * TNFi agents (including, infliximab, adalimumab, certolizumab pegol or golimumab) within 8 weeks prior to randomisation
  * Etanercept within 4 weeks prior to randomisation
  * Leflunomide without cholestyramine wash-out within 8 weeks prior to randomisation
  * Systemic non-biologic medications for PsA or PsO (including traditional Disease-Modifying Antirheumatic Drugs (DMARDs) apremilast, a Janus Kinase (JAK) inhibitor or leflunomide with cholestyramine wash-out) or photochemotherapy within 4 weeks prior to randomisation
  * Intraarticular injections (including steroids) and intramuscular or intravenous corticosteroid treatment within 4 weeks prior to randomisation
  * Topical PsO medications and phototherapy within 2 weeks prior to randomisation
  * Low and high potency opioid analgesics (e.g. tramadol, methadone, hydromorphone, morphine) within 2 weeks prior to randomisation
* Live vaccination ≤ 12 weeks prior to randomisation, or any plan to receive a live vaccination during the conduct of this study. Bacillus Calmette-Guérin (BCG) vaccination is restricted 1 year prior to randomisation through EOO visit.
* further exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-02 (Estimated); Primary Completion 2023-06-26 (Estimated); Study Completion 2023-09-25 (Estimated)

PRIMARY OUTCOMES:
American College of Rheumatology (ACR) 20 response at week 12 | at week 12
  ACR 20 is a binary outcome (Yes, No) with 'yes' indicating improvements of the symptoms.

SECONDARY OUTCOMES:
ACR 50 response at Week 12 | at week 12
  ACR 50 is a binary outcome (Yes, No) with 'yes' indicating improvements of the symptoms.
ACR 70 response at Week 12 | at week 12
  ACR 70 is a binary outcome (Yes, No) with 'yes' indicating improvements of the symptoms.
Change in Tender Joint Count at Week 12 as compared to baseline | at week 12
  Change in Tender Joint Count at Week 12 as compared to baseline, with a maximum possible range between -68 to 68 with higher values indicating a worsening of the symptoms.
Change in Swollen Joint Count at Week 12 as compared to baseline | at week 12
  Change in Swollen Joint Count at Week 12 as compared to baseline, with a maximum possible range between -66 to 66 with higher values indicating a worsening of the symptoms.
Change in Health Assessment Questionnaire-Disability Index (HAQ-DI) at Week 12 as compared to baseline | at week 12
  HAQ-DI score as compared to baseline with a maximum possible range between -3 and 3 with higher values indicating a worsening of the symptoms.
Psoriasis Area and Severity Index (PASI)75 response at Week 12, assessed in patients with a ≥ 3% baseline Psoriasis (PsO) Body Surface Area (BSA) | at week 12
  PASI75 is a binary outcome (Yes, No) with 'Yes' indicating improvements of the symptoms.
Adverse Events | up to 14 weeks
Treatment Emergent Adverse Events | up to 14 weeks
Serious Adverse Events | up to 14 weeks
Intensity of Adverse Events | up to 14 weeks
  Intensity of adverse events will be assessed by Rheumatology Common Toxicity Criteria (RCTC) version 2.0.
  The RCTC criteria consist of 4 grades (1 = mild to 4 = life-threatening) with higher grades indicating a worsening of the symptoms.

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com/